CLINICAL TRIAL: NCT02946125
Title: A Single-Center, Open-Label, Observer-Masked, Active-Controlled, Phase 2 Study of the Safety, Efficacy and Pharmacokinetics of EYN-1601 in Dilation of the Pupil
Brief Title: Study of the Safety, Efficacy and PK of EYN-1601 in Dilation of the Pupil
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eyenovia Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EYN-1601-101
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Mydriasis
MeSH Terms: conditions — Mydriasis | interventions — Phenylephrine; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- MDD-administered EYN-1601 (Experimental): EYN-1601 Ophthalmic Solution administered using the Eyenovia MDD
  Interventions: Combination Product: MDD-administered EYN-1601
- Phenylephrine 2.5% Eyedrop (Active Comparator): Phenylephrine Hydrochloride Ophthalmic Solution 2.5% administered as an eyedrop
  Interventions: Drug: Phenylephrine 2.5% Eyedrop
- Phenylephrine 10% Eyedrop (Active Comparator): Phenylephrine Hydrochloride Ophthalmic Solution 10% administered as an eyedrop
  Interventions: Drug: Phenylephrine 10% Eyedrop

INTERVENTIONS:
Combination Product: MDD-administered EYN-1601 — Phenylephrine hydrochloride ophthalmic solution 10% formulated for microdose spray delivery
  Other Names: MiDD-administered phenylephrine hydrochloride 10%
  Arms: MDD-administered EYN-1601
Drug: Phenylephrine 2.5% Eyedrop — Phenylephrine hydrochloride ophthalmic solution 2.5% eyedrop
  Arms: Phenylephrine 2.5% Eyedrop
Drug: Phenylephrine 10% Eyedrop — Phenylephrine hydrochloride ophthalmic solution 10% eyedrop
  Arms: Phenylephrine 10% Eyedrop

SUMMARY:
This is a Phase 2 study to investigate the safety, efficacy and pharmacokinetics of EYN-1601 for dilation of the pupil. A single microdose of EYN-1601 will be compared to single doses of commercially available phenylephrine hydrochloride 2.5% and 10% ophthalmic solutions.

DETAILED DESCRIPTION:
EYN-1601 delivered topically as a microdose via a proprietary delivery system (the Eyenovia Multi-Dose Device [MDD] system) is being investigated for dilation of the pupil for ophthalmic examinations and procedures. Phenylephrine hydrochloride, a sympathetic α1-adrenergic agonist, has been used for pupil dilation for over 70 years. The mydriatic action of phenylephrine is due to its stimulation of the α1 receptors of the radial muscle of the iris, which causes the muscle fibers to contract and results in pupil dilation.

When conducting a variety of ophthalmological procedures, it is necessary to dilate (enlarge) the pupil to allow an unobstructed view of the lens and retina, as well as the optic nerve. The degree of pupil dilation required is somewhat dependent on the procedure being performed. Eyenovia, the Sponsor, is a specialty pharmaceutical company focused on the development of ophthalmic drug products that can be delivered in small volumes, ie, via microdosing, in order to maximize therapeutic control and minimize systemic absorption. To achieve this goal, Eyenovia is developing a drug/device combination product to allow accurate topical ocular delivery of controlled quantities of specific active pharmaceutical ingredients.

Phenylephrine has been known to cause systemic cardiovascular effects in some patients when dosed via the topical ocular route including hypertension, tachycardia, and more rarely, arrhythmia and stroke, especially in those patients with pre-existing heart conditions. These risks are even more relevant when phenylephrine hydrochloride ophthalmic solution 10% is used in circumstances where a greater degree of mydriasis is required. Microdosing with the Eyenovia MDD system is expected to significantly reduce or eliminate these risks while allowing the same degree of mydriasis produced with the currently approved products.

Subjects (healthy volunteers) will be screened for eligibility and 12 subjects that meet inclusion/exclusion criteria will be enrolled into the study. All subjects will be followed through the same pre-specified treatment visit schedule at which the 3 study drugs are administered (phenylephrine 2.5% eyedrops at Visit 1, phenylephrine 10% eyedrops at Visit 2 and EYN-1601 MDD at Visit 3). At each treatment visit, baseline measurements will be taken prior to study medication administration.

Subjects will participate in safety, efficacy, and pharmacokinetic assessments. Subsequent visits must be separated by at least 2 days but may be up to 1 week apart.

Efficacy will be assessed by measurement of pupil dilation in both eyes.

Safety assessments will include slit lamp examination (SLE) of both eyes and measurement of vital signs (blood pressure [BP]/heart rate [HR]) and adverse events, as well as an ocular discomfort survey

Absorption will be assessed through blood plasma analysis to detect free phenylephrine.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects must be 1-year postmenopausal, surgically sterilized, or women of childbearing potential with a negative urine pregnancy test at Visit 1.
* Provide signed written consent prior to participation in any study-related procedures

Exclusion Criteria:

* Pregnancy or lactation.
* History of diabetes.
* History of cardiac, renal, or hepatic impairment or disease.
* Allergy to phenylephrine hydrochloride.
* Allergy to benzalkonium chloride.
* History of closed-angle glaucoma.
* Anatomically narrow anterior chamber angles (or Shaffer gonioscopic grade of ≥ 2 in either eye).
* Hypertension or treatment for systemic hypertension.
* Ocular surgery or laser treatment of any kind in the study eye within 3 months.
* History of benign prostatic hyperplasia.
* History of chronic or acute uveitis.
* History of traumatic iritis or hyphema.
* History of traumatic mydriasis or angle recession.
* History of anxiety or panic disorders.
* History of thyrotoxicosis, hypothyroidism, or endocrine disease.
* Use of calcium channel blockers, angiotensin-converting enzyme (ACE) inhibitors, benzodiazepines, monoamine oxidase inhibitors, tricyclic antidepressants, anticonvulsants, and systemic steroids (topical, inhaled, intranasal, or perianal steroids are permitted) during the study period.
* Participation in any study of an investigational product or device within 30 days prior to Screening or at any time during the study period.
* Irregularly-shaped pupil secondary to ocular trauma, intraocular surgery or congenital defect.
* History of neurogenic pupil disorder (eg, Horner's syndrome, third cranial nerve palsy, Adie's pupil, Argyl Robertson syndrome, etc.).
* History of anterior chamber intraocular lens (IOL) or iris-fixated IOL.
* History of iris surgery of any kind (eg, iridotomy, iridectomy, coreoplasty)
* History of iris atrophy
* Unwilling to discontinue use of contact lenses on the day of a treatment visit.
* Current active eye disease other than dry eye disease (ie, any disease for which topical or systemic ophthalmic medication is necessary).
* Use of any ophthalmic medication except unpreserved artificial tears on the day of a treatment visit.
* Has a severe/serious ocular condition, or any other unstable medical condition that, in the Investigator's opinion, may preclude study treatment or follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Pupil Dilation | 15, 30, 45, 60, 75, 120 and 180 minutes post administration of study drug
  Mean change in pupil diameter from baseline (prior to study drug administration)

SECONDARY OUTCOMES:
Blood Pressure | 10, 15, 30, 45 and 60 minutes post administration of study drug
  Mean change in blood pressure from baseline (prior to study drug administration)
Heart Rate | 10, 15, 30, 45 and 60 minutes post administration of study drug
  Mean change in heart rate from baseline (prior to study drug administration)
PK (Concentration of free phenylephrine in the blood plasma) | 20 minutes post administration of study drug
  Concentration of free phenylephrine in the blood plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Artesia, California, United States

IPD SHARING:
Plan to Share IPD: No